CLINICAL TRIAL: NCT01642888
Title: A Phase III Trial in Subjects Suspected to Have Tuberculosis, Comparing the Diagnostic Performance of C-Tb to QuantiFERON®-TB Gold In-Tube, in Combination With a Double Blind Randomized Split Body Safety Assessment of C-Tb Versus 2 T.U. Tuberculin PPD RT23 SSI (PPD)
Brief Title: A Trial in Subjects Suspected to Have Tuberculosis, Comparing the Diagnostic Performance of C-Tb to QuantiFERON®, in Combination With a Safety Assessment of C-Tb Versus Tuberculin PPD RT23 SSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: TESEC-05; 2011-005078-40 (EudraCT Number)
Record Dates: First submitted 2012-07-05; First posted 2012-07-17 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.1 µg/0.1 mL C-Tb (Experimental): The C-Tb and 2 T.U. Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT and LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: C-Tb
- 2 T.U. Tuberculin PPD RT 23 SSI (Active Comparator): The C-Tb and 2 T.U. Tuberculin PPD RT 23 SSI agents are given concomitantly to each volunteer in the RIGHT and LEFT forearms according to a double blind randomisation scheme
  Interventions: Biological: 2 T.U. Tuberculin PPD RT 23 SSI

INTERVENTIONS:
Biological: C-Tb — The C-Tb agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Arms: 0.1 µg/0.1 mL C-Tb
Biological: 2 T.U. Tuberculin PPD RT 23 SSI — The 2 T.U. Tuberculin PPD RT 23 SSI agent is administered by the Mantoux injection technique to each volunteer in the RIGHT or LEFT forearm according to a double blind randomisation scheme
  Arms: 2 T.U. Tuberculin PPD RT 23 SSI

SUMMARY:
Tuberculosis (TB) continues to be one of the most serious bacterial infections worldwide and therefore new improved diagnostic tests are needed to help doctors in diagnosing TB.

The new skin test is named C-Tb. Like the current tuberculin skin test, PPD, the C-Tb test is injected just under the skin and will, when positive, show redness and/or swelling at the injection site while a negative test will leave no reactions. The investigators hope that this new C-Tb skin test will be more precise (specific) than the PPD test, as the PPD test e.g. may show a reaction if the person tested is BCG vaccinated.

The aim of this trial is to test the C-Tb skin test in volunteers suspected of having TB disease.

With focus on age, HIV status and CD4 count the following analyses are done (in an overall perspective):

* To compare the C-Tb test to a blood test, the QuantiFERON test.
* To compare the C-Tb test to the PPD test that is currently being used.
* To assess the safety of the C-Tb test.

DETAILED DESCRIPTION:
The TESEC-05 trial is an open comparison of the diagnostics performance of C-Tb compared to the QuantiFERON®-TB Gold In-Tube, in combination with a double-blind randomized split-body safety assessment of C-Tb versus to 2 T.U. Tuberculin PPD RT23 SSI.

The trial is a multi-centre Phase III clinical trial designed specifically to address C-Tb in relation to the paediatric population and to HIV infection. The intention is to evaluate how the C-Tb test performs in the paediatric population with respect to safety, and to ensure that SSI will be able to extrapolate data obtained in an adult population to the paediatric population.

Furthermore, the intention is both to evaluate the diagnostic performance and safety of C-Tb in HIV infected individuals and to evaluate whether SSI will be able to extrapolate data obtained in a non-HIV population to a HIV population.

The trial population will consist of paediatric participants with suspected TB infection and adult participants suspected to have TB disease. Furthermore a control group of 100 children between 5 - 11 years of age with no symptoms or known exposure will be recruited from an area with a "low" prevalence of TB (an area with an incidence rate < 299/100,000 per year, the average rate of TB in South Africa in 2005 was 645/100,000 per year.

The trial will be conducted in South Africa where the prevalence of HIV infection is high and MTb infections are endemic.

BCG vaccination at birth has been common practice since 1961 in South Africa. Thus most of the participants are presumed BCG vaccinated.

ELIGIBILITY:
Inclusion Criteria:

HIV NEGATIVE PARTICIPANTS:

1. Participants between 5 and 65 years attending the TB clinic due to suspicion of TB disease
2. Infants, toddlers and children between 28 days and 4 years must either have symptoms or signs of TB or be in close contact to a smear positive pulmonary TB case (more than 6 hours/day for at least five days)
3. Is between 28 days and 65 years of age
4. Participant, parent or legal guardian has signed the informed consent
5. Is HIV negative confirmed by two rapid tests. However, children between 28 days and 4 years may have an unknown HIV status and may receive antiretroviral therapy (ART) or have breastfeeding mothers on ART
6. Is willing and likely to comply with the trial procedures
7. Is prepared to grant authorized persons access to their medical record

HIV POSITIVE PARTICIPANTS:

1. Participants between 5 and 65 years attending the TB clinic due to suspicion of TB disease
2. Infants, toddlers and children between 28 days and 4 years must either have symptoms* or signs** of TB or be in close contact to a smear positive pulmonary TB case (more than 6 hours/day for at least five days)
3. Is between 28 days and 65 years of age
4. Participant, parent or legal guardian has signed the informed consent
5. Is HIV positive confirmed by:

   1. two positive rapid tests or
   2. 1 positive rapid test and an additional confirmatory ELISA test
6. A CD4 count has been done
7. Is willing and likely to comply with the trial procedures
8. Is prepared to grant authorized persons access to their medical record

HIV NEGATIVE CONTROL GROUP:

1. Participant with no known contact to people infected with MTb and no signs or symptoms of TB.
2. Is between 5 and 11 years of age
3. Participant, parent or legal guardian has signed the informed consent
4. Is HIV negative confirmed by two rapid tests
5. Is willing and likely to comply with the trial procedures
6. Is prepared to grant authorized persons access to their medical record

Exclusion Criteria:

HIV NEGATIVE PARTICIPANTS:

1. Has a confirmed diagnosis of tuberculosis at Screening Visit
2. Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. MMR, yellow fever, oral typhoid vaccines) except BCG vaccine
3. Has been tuberculin (TST) tested less than 12 months prior to the day of inclusion
4. Is pregnant, breastfeeding or intending to get pregnant during the trial period
5. Is a female of child bearing potential (12 years of age or older) not willing to use effective barrier (including spermicidal gel), hormonal or intrauterine contraceptive measures during the trial period
6. Has an active disease affecting the lymphoid organs (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
7. Has a current skin condition which interferes with the reading of the C-Tb and PPD e.g. tattoos, severe scarring, burns/sunburns, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
8. Has a condition where blood drawings pose more than minimal risk for the participant, such as haemophilia, other coagulation disorders or significantly impaired venous access
9. Currently participating in another clinical trial with an investigational or non-investigational drug or device or has participated in another clinical trial within the 3 months prior to dosing
10. Has participated in previous clinical trials investigating the ESAT-6 and/or CFP-10 antigens
11. Has a condition which in the opinion of the investigator is not suitable for participation in the trial

HIV POSITIVE PARTICIPANTS:

1. Has a confirmed diagnosis of tuberculosis at Screening Visit
2. Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. MMR, yellow fever, oral typhoid vaccines)
3. Has been tuberculin (TST) tested less than 12 months prior to the day of inclusion
4. Is pregnant, breastfeeding or intending to get pregnant during the trial period
5. Is a female of child bearing potential (12 years of age or older) not willing to use effective barrier (including spermicidal gel), hormonal or intrauterine contraceptive measures during the trial period
6. Has an active disease affecting the lymphoid organs except for HIV (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
7. Has a known diagnosis of AIDS or is receiving antiviral therapy at the time of Screening Visit
8. Has a current skin condition which interferes with the reading of the C-Tb and PPD e.g. tattoos, severe scarring, burns/sunburns, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
9. Has a condition where blood drawings pose more than minimal risk for the participant, such as haemophilia, other coagulation disorders or significantly impaired venous access
10. Currently participating in another clinical trial with an investigational or non-investigational drug or device or has participated in another clinical trial within the 3 months prior to dosing
11. Has participated in previous clinical trials investigating the ESAT-6 and/or CFP-10 antigens
12. Has a condition which in the opinion of the investigator is not suitable for participation in the trial

HIV NEGATIVE CONTROL GROUP:

1. Has been vaccinated with a live vaccine within 6 weeks prior to the day of inclusion (e.g. MMR, yellow fever, oral typhoid vaccines) except BCG vaccine
2. Has been tuberculin (TST) tested less than 12 months prior to the day of inclusion
3. Has an active disease affecting the lymphoid organs (e.g., Hodgkin's disease, lymphoma, leukaemia, sarcoidosis)
4. Has a current skin condition which interferes with the reading of the C-Tb and PPD e.g. tattoos, severe scarring, burns/sunburns, rash, eczema, psoriasis, or any other skin disease at or near the injection sites
5. Has a condition where blood drawings pose more than minimal risk for the participant, such as haemophilia, other coagulation disorders, or significantly impaired venous access
6. Currently participating in another clinical trial with an investigational or non-investigational drug or device, or has participated in another clinical trial within the 3 months prior to dosing
7. Has participated in previous clinical trials investigating the ESAT-6 and/or CFP-10 antigens
8. Has a condition which in the opinion of the investigator is not suitable for participation in the trial

Ages: 28 Days to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1190 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of C-Tb in relation to age, HIV and CD4 counts | Onset between the injections and 28 days after the injections
To evaluate the clinical safety of C-Tb, with emphasis on children and HIV positive participants | Onset between the injections and 28 days after the injections

SECONDARY OUTCOMES:
To evaluate the difference in sensitivity between C-Tb and QuantiFERON®-TB Gold in-Tube in trial participants with confirmed TB diagnosis, overall, and according to age and HIV status. | From injections to 2-3 days after the injections
To evaluate the difference in sensitivity between C-Tb and Tuberculin PPD RT23 SSI in trial participants with confirmed TB diagnosis overall, and according to age and HIV status. | Onset between the injections and 28 days after the injections
To evaluate the difference in specificity between C-Tb and QuantiFERON®-TB Gold in-Tube in the control group of 100 children aged 5 - 11 years with no TB symptoms and no known exposure to MTb overall, and according to age. | From injections to 2-3 days after the injections
To evaluate the difference in specificity between C-Tb and Tuberculin PPD RT23 SSI in the control group of 100 children aged 5 - 11 years with no TB symptoms and no known exposure to MTb overall, and according to age. | Onset between the injections and 28 days after the injections
To compare the diagnostic outcome of C-Tb to that of QuantiFERON®-TB Gold in-Tube using a latent class approach | From injections to 2-3 days after the injections
To compare the diagnostic outcome of C-Tb to that of Tuberculin PPD RT23 SSI using a latent class approach | Onset between the injections and 28 days after the injections
To evaluate the diagnostic performance of Tuberculin PPD RT23 SSI in relation to age, HIV status and CD4 counts | Onset between the injections and 28 days after the injections
To evaluate the clinical safety of Tuberculin PPD RT23 SSI | Onset between the injections and 28 days after the injections
To evaluate the diagnostic performance of QuantiFERON®-TB Gold in-Tube in relation to age, HIV status and CD4 counts | On the day of the injections

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Diacon, MD, Principal Investigator — M2 Karl Bremer Hospital; Henrik Aggerbeck, M.Sc., Study Chair — Statens Serum Institut
Locations (9):
- South Africa (9):
  - Primecure Medicentre, Mercantile Hospital, Port Elizabeth, Eastern Cape
  - Worthwhile Clinical Trials, Lakeview Hospital, Benoni, Gauteng
  - Synnyside Medi-Clinic, Pretoria, Gauteng
  - Synexus Stanza Bopape Clinic, Pretoria, Gauteng
  - Setshaba Research Centre, Pretoria, Gauteng
  - M2 Karl Bremer Hospital, Bellville, Cape Town, Western Cape
  - Tiervlei Trial Centre, Karl Bremer Hospital, Bellville, Cape Town, Western Cape
  - UCT Lung Institute, Groote Schuur Hospital, Cape Town, Western Cape
  - Be Part Yoluntu Centre, Paarl, Western Cape

REFERENCES:
- [Derived] Aggerbeck H, Ruhwald M, Hoff ST, Borregaard B, Hellstrom E, Malahleha M, Siebert M, Gani M, Seopela V, Diacon A, Lourens M, Andersen P, Dheda K. C-Tb skin test to diagnose Mycobacterium tuberculosis infection in children and HIV-infected adults: A phase 3 trial. PLoS One. 2018 Sep 24;13(9):e0204554. doi: 10.1371/journal.pone.0204554. eCollection 2018. PMID 30248152